CLINICAL TRIAL: NCT03695146
Title: Heart Inflammation and Mental Stress Study
Acronym: HIMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Roger McIntosh, Assistant Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 20180631; K01HL139722-01 (NIH)
Record Dates: First submitted 2018-09-28; First posted 2018-10-03 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Hypertension
Keywords: High blood pressure; HIV
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Paced breathing (Experimental): Individuals will be asked to sit in a quiet room while sensors collect their heart rate, respiratory rate and blood pressure for approximately 45 minutes. Individuals in this arm will engage in a paced breathing. Initial respiratory rate will be measured with a transducer. Participants will be connected to a paced breathing device (RESPERATE) that will gradually reduce the pace of audio tones presented to those individuals from spontaneous breathing rate down to 6 - 8 breaths per minute.
  Interventions: Behavioral: Paced breathing
- Relaxing music (Active Comparator): Individuals will be asked to sit in a quiet room while sensors collect their heart rate, respiratory rate and blood pressure for approximately 45 minutes. Individuals will be provided with an audio device that plays soothing/relaxing music at a similar range (beats per minute) of the auditory signal presented during the experimental condition. Subjects will not be instructed how to breathe in this arm.
  Interventions: Behavioral: Active relaxation
- No intervention (No Intervention): Individuals will be asked to sit in a quiet room while sensors collect their heart rate, respiratory rate and blood pressure for approximately 45 minutes.

INTERVENTIONS:
Behavioral: Paced breathing — Individuals will be fitted with a respiratory transducer and receive auditory tones with which to pace their rate of inspiration and expiration in the experimental group.
  Arms: Paced breathing
Behavioral: Active relaxation — Individuals will be provided with headphones while resting quietly listening to relaxing tones/music.
  Arms: Relaxing music

SUMMARY:
The aim of the study is to investigate the neural underpinnings of cardiovascular reactivity to mental stress as a function of HIV and hypertensive risk.

DETAILED DESCRIPTION:
The main objectives of the study are to assess (1) patterns of brain activity/connectivity that confers greater cardio-autonomic/emotion regulation, (e.g., heart rate variability, blood pressure reactivity, inflammatory-immune activation, etc.), during rest, mental stress, and anger-related distress, (2) whether changes in breathing pace mitigate task-based effects on cardio-autonomic-immune regulation, and (3) whether these patterns vary as a function of HIV or pre-hypertensive (HTN) status-related changes to the brain structures underlying cardioautonomic and emotion regulation.

ELIGIBILITY:
Inclusion criteria:

1. pre-hypertension screening.
2. HIV-antibody testing.

Exclusion criteria:

1. current use of anti-lipid, antihypertensive, or heart rate altering medications;
2. current or lifetime history of cardiovascular disease diagnosis or treatment including pulmonary stenosis, heart valve abnormalities and hypertension;
3. current or lifetime diagnoses of cancer, kidney/liver disease, hypertension, Type 1 or Type 2 diabetes;
4. history of trauma, cerebral infarction or hemorrhage;
5. current diagnosis and/or treatment for hypertension;
6. severe cognitive impairment;
7. current treatment or diagnosis of psychiatric illness;
8. metal implants or debris within the body; or pregnancy;
9. body mass index > 35;
10. use of hormone replacement therapy; and current smoker.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-08-19 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-22 (Actual)

PRIMARY OUTCOMES:
Change in heart rate variability | Baseline, pre-intervention and up to 60 minutes post-intervention
  Heart rate variability will be measured using a standard electrocardiogram to detect variability in R -to-R intervals.

SECONDARY OUTCOMES:
Change in cytokine expression in peripheral blood mononuclear cells | Baseline, pre-intervention and up to 60 minutes post-intervention
  Peripheral blood will be drawn and mononuclear cells isolated and incubated with lipopolysaccharide to induce inflammatory cytokine expression. The change in cytokine expression will be quantified as a function of time.

CONTACTS AND LOCATIONS:
Overall Officials: Roger C McIntosh, Ph.D., Principal Investigator — University of Miami, College of Arts and Sciences
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No